CLINICAL TRIAL: NCT02584998
Title: Reducing Colorectal Cancer Death Through Mailed Outreach Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PPO 14-369; 01522 (Other: Corporal Michael J. Crescenz VA Medical Center)
Record Dates: First submitted 2015-10-21; First posted 2015-10-23 (Estimated); Results first posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual care (No Intervention): These patients will continue to receive the current practice at the Philadelphia VA Medical Center (VAMC) of offering screening during an office visit. Other interventions will be embedded within this existing program for a pragmatic approach. However, all participants in the trial, including those in usual care (UC), will receive follow-up of test results and navigation to diagnostic colonoscopy for positive FIT results.
- Screening invitation-reminder (Active Comparator): Participants will receive UC and also receive an invitation letter with information about CRC testing. The information will include lay-audience description of screening tests and symptoms that should prompt diagnostic work-up. The packet will have instructions to contact the study team if participants believe they are not eligible and to update the contact information on record. The letter will inform participants that a telephone reminder will follow in 4 weeks from invitation letter if screening is not completed. They will also receive notification of test results and navigation to colonoscopy, if needed. For the purposes of this intervention, Week 1 will be the week the invitation letter was sent (time zero).
  Interventions: Other: Screening invitation-reminder
- Mailed-FIT (Active Comparator): Participants randomized to Mailed-FIT will receive a mailed FIT pre-notification letter (plus a screening invitation) followed by the kit 1 week later. Participants will receive instructions to contact the study team if they believe they are not eligible and to update their contact information. They will be informed that a telephone reminder will follow 4 weeks from notification letter if screening is not completed. Participants who do not return their kit within 4 weeks after their pre-notification letter was mailed will receive a live telephone reminder, followed by 2 additional calls at the end of weeks 5 and 6, if needed. For the purposes of this intervention, Week 1 will be the week the pre-notification letter was sent (time zero).
  Interventions: Other: Mailed-FIT

INTERVENTIONS:
Other: Mailed-FIT — The FIT is analyzed at the Philadelphia VAMC by an auto-analyzer system that provides quantitative results corresponding to the concentration of hemoglobin in the collected sample. Specimens will be analyzed according to manufacturer's instructions to minimize potential degradation of hemoglobin. Results are provided as positive if the hemoglobin concentration is 100ng/dL. The machine records (but does not report) the quantitative results of the hemoglobin concentration in the sample, which we will seek to obtain from the laboratory for future studies.
  Other Names: Fecal Immunochemical Test
  Arms: Mailed-FIT
Other: Screening invitation-reminder — These patients will continue to receive UC. They will in addition receive an invitation letter with all of the information about CRC testing in the mail-FIT arm
  Arms: Screening invitation-reminder

SUMMARY:
The main study aim is to develop, implement and disseminate a pilot population-based mailed FIT outreach screening program in the Philadelphia VA Medical Center that does not rely on having an office visit, by conducting a proof-of-concept 3-arm parallel-design pragmatic randomized trial to (1) Compare the effects of usual care (UC), screening invitation + reminder (invitation-reminder), or screening invitation + mailed FIT kit + reminder (mailed-FIT); (2) Explore whether the FIT completion rate varies by age or race/ethnicity; and (3) Explore barriers to use of mailed outreach screening for Veterans.

DETAILED DESCRIPTION:
This study seeks to establish the foundation to systematically study and improve the delivery and effectiveness of colorectal cancer (CRC) screening in the VA by developing, implementing and disseminating a pilot mailed-FIT screening outreach program that does not rely on having a clinical office visit. The investigators specifically address the need to identify and remediate potential failures to identify and offer screening to eligible Veterans through multilevel interventions. The investigators will also create electronic data linkages to, in future studies, enable evaluation of FIT performance characteristics and help close critical evidence gaps for optimizing screening among Veterans. As this is a pilot study, the focus is to assess feasibility of a population-based screening outreach approach through the development, implementation and dissemination of a mailed FIT outreach program in the Philadelphia VA Medical Center that does not rely on having an office visit.

ELIGIBILITY:
Inclusion Criteria:

* The pragmatic trial will include Veterans in southeastern Pennsylvania and Southern New Jersey who, during the funding year
* 50 to 75 years old
* Have received care at the Philadelphia VA Medical Center in the 18-48 months prior to selection for the study but who have not been seen by primary care in the past 18 months prior to selection
* Due for screening
* Are asymptomatic for CRC
* This includes the period during which 3-sample testing was being regularly used at the Philadelphia VA Medical Center

Exclusion Criteria:

* Have any known gastrointestinal symptoms such as:

  * bleeding
  * unexplained weight loss
  * change in bowel habits
  * family history of CRC
  * inflammatory bowel disease (IBD)
  * colectomy using International Classification of Disease (9th and 10th edition) diagnostic code or by self-report.
* The investigators will also exclude Veterans:

  * with evidence of prior colonoscopy within 10 years
  * sigmoidoscopy within 5 years
  * fecal occult blood test (FOBT)/FIT in the same calendar year
* The information used to exclude patients will be derived from the electronic queries or chart audits.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 782 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Carter Paulson, MD MSCE, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldshore MA, Mehta SJ, Fletcher W, Tzanis G, Doubeni CA, Paulson EC. An RCT of Fecal Immunochemical Test Colorectal Cancer Screening in Veterans Without Recent Primary Care. Am J Prev Med. 2020 Jul;59(1):41-48. doi: 10.1016/j.amepre.2020.02.014. PMID 32564804

RESULTS

PARTICIPANT FLOW:
Groups:
- Mailed-FIT: Participants randomized to Mailed-FIT will receive a mailed FIT pre-notification letter (+screening invitation) followed by kit 1 week later. Participants will receive instructions to contact the study team if they believe they are not eligible and to update contact information. They will be informed that a telephone reminder will follow 4 weeks from letter if screening not completed. Participants who do not return their kit in 4 weeks will receive a telephone reminder, followed by 2 additional calls at the end of weeks 5 and 6, if needed. For the purposes of this intervention, Week 1 will be the week the pre-notification letter was sent (time zero).
  Mailed-FIT: The FIT is analyzed at the Philadelphia VAMC by an auto-analyzer system that provides quantitative results corresponding to the concentration of hemoglobin in the collected sample.
Period: Overall Study
Arm/Group | Usual Care | Screening Invitation-reminder | Mailed-FIT
Started | 260 | 261 | 261
Completed | 260 | 261 | 261
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Screening Invitation-reminder | Mailed-FIT | Total
Number analyzed (Participants) | 260 | 261 | 261 | 782
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (7.0) | 60 (7.0) | 61 (6.5) | 61 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 7 | 22
  Male | 252 | 254 | 254 | 760
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 162 | 149 | 160 | 471
  Race: White | 85 | 97 | 88 | 270
  Race: Other | 3 | 4 | 5 | 12
  Race: Unknown | 10 | 11 | 8 | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 260 | 261 | 261 | 782

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Completed the Mailed FIT Test Screening Within 6 Months
Description: The completion rate of mailed FIT test within 6 months of the mailing of the screening invitation. The absence of FIT result in the electronic medical record (CRPS) will be considered a failure to complete the FIT test
Time Frame: 6 months
Population: For this outcome, we just analyzed patients in Arm 3 (n=261), the mailed-FIT kit, arm, as they were the only patients eligible to return a mailed fit kit.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Screening Invitation-reminder | Mailed-FIT
Number analyzed (Participants) | 0 | 0 | 261
Participants | 0 | 0 | 62

2. Secondary Outcome: The Number of Participants Who Received Any Colorectal Cancer Screening Test in the 6-month Period After Enrollment Into the Study.
Description: The receipt of any colorectal cancer screening test in the 6-month period after enrollment into the study. For patients in the usual care arm, 6 months was counted from the date of mailed letter to arms 2 and 3 within that block of participants.
Time Frame: 6 months
Population: We analyzed all randomized patients to identify any CRC screening at 6 months from mailed screening invitation.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Screening Invitation-reminder | Mailed-FIT
Number analyzed (Participants) | 260 | 261 | 261
Participants | 15 | 20 | 68
Statistical Analysis 1: Comparison: Usual Care vs Screening Invitation-reminder vs Mailed-FIT; In our power and sample size analysis, we assumed 15% screening rate in usual care, 25% with invitation, and 40% with mailed-FIT. A sample size of 500 (250/arm) will give 80% power for UC vs. screening invitation-reminder, and 152/arm will give a power of 80% for the screening invitation-reminder vs. mailed-FIT. Accounting for the possibility that up to 20% of participants could be ineligible post-randomization, we concluded that we should enroll 783 patients, 261 per arm, for this trial; Test type: Other; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the same time frame as the primary outcome, which was 6 months from the time of the mailed screening invitation in arms 2 and 3.
Arm/Group | Usual Care | Screening Invitation-reminder | Mailed-FIT
All-Cause Mortality (participants affected / at risk) | 1/260 | 0/261 | 0/261
Serious Adverse Events (participants affected / at risk) | 0/260 | 0/261 | 0/261
Other Adverse Events (participants affected / at risk) | 0/260 | 0/261 | 0/261

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT02584998/Prot_SAP_000.pdf